CLINICAL TRIAL: NCT06421792
Title: Scanning Electron Microscopy (SEM) and Confocal Imaging of Clot in Two Different Protamine Environments (PrOtamIne doSing clOt imagiNg (POISON) Study)
Brief Title: PrOtamIne doSing clOt imagiNg (POISON) Study
Acronym: POISON
Status: Not yet recruiting | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: University of Oxford (Other); University of Liverpool (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: T03024
Record Dates: First submitted 2024-04-21; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard: 10 patients receiving standard reversal with 1:1 protamine / heparin ratio
- PRODOSE Algorithm: 10 patients who had heparin reversed using the PRODOSE algorithm anticipated (average protamine / heparin ratio 0.6:1).

SUMMARY:
The proposed study involves using two different high-resolution microscopic imaging techniques to examine the health and platelet invasion of clot in patients who were given 1:1 protamine / heparin and compare this to clot from patients who had heparin reversed using the PRODOSE algorithm. Patients will be treated according to the routine clinical practice of their individual care team.

DETAILED DESCRIPTION:
Sample collection at RPH

Patients will have a total of 14ml of blood taken during the procedure.

The first 7ml will be taken after induction of anaesthesia along with routine blood gas and coagulation sampling through the routinely indwelling arterial catheter. The initial sample must be taken before any heparin has been administered. This will be used to fill 2 x 3.5ml citrated (green top) blood tubes. These will be clearly labelled as "pre-heparin" with a Tissue Bank ID number.

The second 7ml will be taken 5 minutes after heparin has been reversed with protamine after cessation of cardiopulmonary bypass. It will again be taken at the same time as routine sampling for blood gas and coagulation studies. Analog to the first sample, it will again be divided and used to fill 2 x 3.5ml citrated (green top) blood tubes. These will be clearly labelled as "post-protamine" with the same ID number and whether "1:1" or a "PRODOSE algorithm determined" protamine: heparin ratio was used.

In keeping with clinical routine, ROTEM coagulation testing and full blood counts will be requested as seen necessary by the clinical team.

The samples will be sent to Royal Papworth Hospital (RPH) Tissue Bank for initial processing. Samples need to be processed within 4 hours of blood draw.

After initial processing, samples will be sent for confocal imaging to the MRC Laboratory of Molecular Biology (LMB) and for SEM imaging to the University of Oxford respectively.

Clinical data to be collected (to be completed by anaesthetic team).

1. Demographic information: Age / Gender / Weight / Height / Medication history;
2. Type of surgery;
3. Cardiac drug history and antiplatelets / anticoagulants and timing;
4. Coagulation tests (ACT / ROTEM) at the following points: a) Pre-heparin, b) Post-heparin, pre-CPB, c) Throughout CPB, c) Post-protamine;
5. Full blood count at the following points: a) Pre-surgery and date of sample, b) Post-protamine; 6) CPB and x-clamp times, nadir temperature

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective, uncomplicated single procedure cardiac surgery with anticipated CPB duration < 120 min
* with all anticoagulant drugs stopped at least 5 days before surgery, apart from aspirin
* with normal full blood count and clotting screen pre-OP.

Exclusion Criteria:

* emergency surgery
* inability to stop anticoagulants except aspirin for 5 days pre-OP
* complex surgery with anticipated CPB duration > 120min
* operations planned to be done at temperature on CPB < 34 degrees
* operations requiring deep hypothermic circulatory arrest, solid organ transplantation
* know blood dyscrasia
* intra-operative blood or blood product transfusion or post-operative coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective, uncomplicated single procedure cardiac surgery with anticipated CPB duration < 120 min
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-08 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
High-resolution microscopic images (Scanning Electron Microscopy and Confocal Imaging) | Pre Heparin and Post Protamine [5 minutes after heparin has been reversed]
  The proposed study involves using two different high-resolution microscopic imaging techniques to examine the health and platelet invasion of clot in patients who were given 1:1 protamine / heparin and compare this to clot from patients who had heparin reversed using the PRODOSE algorithm.
  This is an observational study in which differences between images of clot obtained from samples from the two patient groups and before and after cardiopulmonary bypass will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Small observational study so IPD not relevant

REFERENCES:
- [Background] Miles LF, Burt C, Arrowsmith J, McKie MA, Villar SS, Govender P, Shaylor R, Tan Z, De Silva R, Falter F. Optimal protamine dosing after cardiopulmonary bypass: The PRODOSE adaptive randomised controlled trial. PLoS Med. 2021 Jun 7;18(6):e1003658. doi: 10.1371/journal.pmed.1003658. eCollection 2021 Jun. PMID 34097705